CLINICAL TRIAL: NCT05735795
Title: Feasibility of Carbon Dye Marking of Axillary Lymph Nodes Before Neoadjuvant Chemotherapy in Patients With Breast Cancer
Brief Title: Feasibility of Carbon-Dye Marking of Axillary Lymph Nodes Before Neoadjuvant Chemotherapy in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Yıldırım, Assoc. Prof., Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-09
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; Lymph node metastasis; Targeted axillary dissection; Nodal marking
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carbon Black Tattoo arm (Other): In patients with breast cancer diagnosed with positive axillary lymph node involvement by fine needle aspiration cytology, 0.1-0.5 ml Carbon Black Tattoo dye will be applied simultaneously to the lymph node capsule and surrounding tissue, while clips are placed on the axilla before starting neoadjuvant chemotherapy. After the neoadjuvant treatment is completed, the patient who is taken into surgery will be injected with periareolar blue dye as in the standard practice, and blue stained node, clipped node and carbon stained node will be searched as sentinal lymph node. The removed lymph nodes will be evaluated histopathologically in terms of metastasis with a frozen study during the operation, and if metastasis is detected, axillary lymph node dissection will be performed
  Interventions: Other: Carbon Black Tattoo

INTERVENTIONS:
Other: Carbon Black Tattoo — SPOT ENDOSCOPIC MARKER is an FDA (American Food and Drug Administration) approved Carbon Black Tattoo paint that has been used for a long time to mark lesions in the gastrointestinal tract.

SUMMARY:
Although treatment is started with surgery in early stage tumors depending on the molecular subtype, neoadjuvant chemotherapy is the initial treatment in locally advanced tumors or if axillary lymph node involvement is present.

Axillary lymph node dissection (ALND) has been used for a very long time in the traditional approach to the treatment of breast cancer. The current approach in patients with early stage, clinically negative breast cancer of the axilla is sentinel lymph node biopsy (SLNB). SLNB is done to evaluate the axilla in both early stage tumors and suitable patients after NAC. According to ACOSOG Z1071, when at least 3 lymph nodes were removed using lymphoscintigraphy and blue dye for SLNB, the false-negative rate was found to be less than 10% in patients with proven axillary involvement, and SLNB was shown to be feasible after NAC. Targeted axillary dissection (TAD) is a procedure that includes SLND with removal of the lymph node identified and marked as containing metastatic disease before treatment. Multiple clinical studies have shown that TAD is a viable option to reduce false-negativeness in patients with breast cancer after NAC. In patients with axillary involvement, a metallic clip is placed in the suspected lymph node prior to neoadjuvant therapy and a radioactive iodine-125 seed is implanted into the target after completion of chemotherapy, and during TAD, the core node is removed using a radioactive probe. Today, the applicability of these procedures is difficult due to both the cost and the absence of nuclear medicine units in some hospitals. For this reason, alternative methods that can be applied more easily in the evaluation of the axilla after NAC are being investigated. SPOT ENDOSCOPIC MARKER is an FDA (American Food and Drug Administration) approved Carbon Black Tattoo paint that has been used for a long time to mark lesions in the gastrointestinal tract. Its shelf life is 20 months. In our project, in patients with lymph node involvement in the axilla who have had a metallic clip placed with biopsy before NAC, the lymph node will be marked with a Spot Endoscopic Marker simultaneously, and the permanence of the spot marker dye will be evaluated by excising the clip-marked and black-painted lymph node in addition to the methylen blue injected during the operation. The reliability of the use of Spot Endoscopic Marker, which is much cheaper instead of clips, for permanent axillary marking in TAD will be evaluated.

DETAILED DESCRIPTION:
Breast cancer affects millions of women worldwide. According to the statistics, 2.3 million new cases of breast cancer were reported in 2020. Although treatment is started with surgery in early stage tumors depending on the molecular subtype, neoadjuvant chemotherapy is the initial treatment in locally advanced tumors or if axillary lymph node involvement is present. With NAC in locally advanced breast cancer, it is possible to both shrink the tumor and make patients who were initially inoperable suitable for surgery, and increase the feasibility of breast-conserving surgery.

Although axillary lymph node dissection (ALND) has been used for a very long time in the traditional approach to the treatment of breast cancer, the current approach in patients with early stage, clinically negative breast cancer of the axilla is sentinel lymph node biopsy (SLNB). SLNB is done to evaluate the axilla in both early stage tumors and suitable patients after NAC. According to ACOSOG Z1071, when at least 3 lymph nodes were removed using lymphoscintigraphy and blue dye for SLNB, the false-negative rate was found to be less than 10% in patients with proven axillary involvement, and SLNB was shown to be feasible after NAC. Targeted axillary dissection (TAD) is a procedure that includes SLND with removal of the lymph node identified and marked as containing metastatic disease before treatment. Multiple clinical studies have shown that TAD is a viable option to reduce false-negativeness in patients with breast cancer after NAC. In patients with axillary involvement, a metallic clip is placed in the suspected lymph node prior to neoadjuvant therapy and a radioactive iodine-125 seed is implanted into the target after completion of chemotherapy, and during TAD, the core node is removed using a radioactive probe. The procedure is performed with SLND using the dual-tracer technique. Today, the applicability of these procedures is difficult due to both the cost and the absence of nuclear medicine units in some hospitals. For this reason, alternative methods that can be applied more easily in the evaluation of the axilla after NAC are being investigated. SPOT ENDOSCOPIC MARKER is an FDA (American Food and Drug Administration) approved Carbon Black Tattoo paint that has been used for a long time to mark lesions in the gastrointestinal tract. Its shelf life is 20 months. In our project, in patients with lymph node involvement in the axilla who have had a metallic clip placed with biopsy before NAC, the lymph node will be marked with a Spot Endoscopic Marker simultaneously, and the permanence of the spot marker dye will be evaluated by excising the clip-marked and black-painted lymph node in addition to the methylen blue injected during the operation. The reliability of the use of Spot Endoscopic Marker, which is much cheaper instead of clips, for permanent axillary marking in TAD will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced breast cancer known to have metastases to the axillary lymph nodes at baseline and referred for neoadjuvant chemotherapy will be included in the study.

Exclusion Criteria:

* diagnosis by excisional biopsy
* previous axillary surgery
* failure to complete neoadjuvant therapy
* progression during therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
The reliability of the use of Spot Endoscopic Marker | 12 months
  Carbon tattoo is an FDA-approved dye that is used to mark lesions in the gastrointestinal tract in vivo. It is used in lesion follow-up because it is permanent for a long time. In current practice, lymph nodes with biopsy-proven axillary lymph node involvement before neoadjuvant chemotherapy are marked with a metallic clip before starting the treatment and excised as sentinal lymph node during surgery. This procedure is both expensive and difficult to implement due to the necessity of having a nuclear medicine department in the hospital. Our aim in this study is to evaluate the excision of the lymph node by marking it with carbon dye instead of a clip.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Yildirim, Assoc. Prof., Principal Investigator — Gaziosmanpasa Training and Research Hospital
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)